CLINICAL TRIAL: NCT03751657
Title: An Investigational Trial Comparing the Efficacy and Safety of Once Weekly NNC0148-0287 C (Insulin 287) Versus Once Daily Insulin Glargine, Both in Combination With Metformin, With or Without DPP-4 Inhibitors, in Insulin naïve Subjects With Type 2 Diabetes Mellitus
Brief Title: A Research Study to Compare Insulin 287 Once a Week to Insulin Glargine (100 Units/mL) Once a Day in People With Type 2 Diabetes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1436-4383; U1111-1208-4124 (Other: World Health Organization (WHO)); 2018-000322-63 (EudraCT Number)
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; Metformin; Dipeptidyl-Peptidase IV Inhibitors; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin 287 (Experimental): Participants will receive once weekly insulin 287 and once daily placebo in combination with metformin with or without dipeptidyl peptidase-4 inhibitors (DPP4i) during 26 weeks of treatment period.
  Interventions: Drug: Insulin icodec; Drug: Metformin; Drug: Dipeptidyl peptidase-4 inhibitors; Drug: Placebo (insulin glargine)
- Insulin glargine (Active Comparator): Participants will receive once daily insulin glargine and once weekly placebo in combination with metformin with or without DPP4i during 26 weeks of treatment period.
  Interventions: Drug: Placebo (insulin 287); Drug: Metformin; Drug: Dipeptidyl peptidase-4 inhibitors; Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin icodec — Insulin 287 once weekly subcutaneous (s.c.) injections at the starting dose of 70 units. Dose adjustment was done for the individual patient based on the three pre-breakfast self-measured plasma glucose values measured on two days prior to titration and on the day of the contact. The insulin dose adjustment should aim to reach an SMPG of 3.9-6.0 mmol/L (70-108 mg/dL)
  Other Names: Insulin 287
  Arms: Insulin 287
Drug: Placebo (insulin 287) — Participants will receive once weekly s.c. injections of placebo equivalent to insulin 287.
  Arms: Insulin glargine
Drug: Metformin — Metformin is considered as non investigational medicinal product. Subject will continue metformin at stable pre-trial dose.
Drug: Dipeptidyl peptidase-4 inhibitors — Dipeptidyl peptidase-4 inhibitors are considered as non investigational medicinal products. Subject will continue dipeptidyl peptidase-4 inhibitor at stable pre-trial dose.
Drug: Insulin glargine — Insulin glargine (100 U/mL) once daily s.c. injections at the starting dose of 10 units. Dose adjustment will be done for the individual patient based on the three pre-breakfast self-measured plasma glucose values measured on two days prior to titration and on the day of the contact. The insulin dose adjustment should aim to reach an SMPG of 3.9-6.0 mmol/L (70-108 mg/dL).
  Arms: Insulin glargine
Drug: Placebo (insulin glargine) — Participants will receive once daily s.c. injections of placebo equivalent to insulin glargine.
  Arms: Insulin 287

SUMMARY:
The study compares 2 medicines for people with type 2 diabetes: insulin 287 (a new medicine) and insulin glargine (a medicine doctors can already prescribe). The study doctors will test insulin 287 to see how well it works compared to insulin glargine. The study will also test if insulin 287 is safe. The study participants will either get insulin 287 or insulin glargine (100 units/mL) - which treatment the participants get is decided by chance. The participants will need to inject their selves every day about the same time. Once a week the participant will need to take 1 extra injection on the same day of the week. The participants will have 16 clinic visits and 14 phone calls with the study doctor. During the study, the doctors will ask you to: 1) measure your blood sugar every day with a blood glucose meter using a finger prick, 2) write down different information in a paper diary daily and return this to your doctor, 3) wear a medical device to measure your blood sugar all the time for 2 weeks 5 times during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days prior to the day of screening
* HbA1c of 7.0-9.5% (53-80 mmol/mol) (both inclusive) as assessed by central laboratory
* Stable daily dose(s) for 90 days prior to the day of screening of any of the following antidiabetic drug(s) or combination regime(s): Any metformin formulations greater than or equal to 1500 mg or maximum tolerated or effective dose (as documented in subject's medical record) OR Any metformin formulations greater than or equal to 1500 mg or maximum tolerated or effective dose (as documented in subject medical record) with Dipeptidyl peptidase-4 inhibitor (DPP4i) (greater than or equal to half of the maximum approved dose according to local label or maximum tolerated or effective dose (as documented in subject's medical records)
* Insulin naïve. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes
* Body mass index (BMI) less than or equal to 40.0 kg/m^2

Exclusion Criteria:

* Any episodes of diabetic ketoacidosis within the past 90 days prior to the day of screening and between screening and randomisation
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening and between screening and randomisation
* Presently classified as being in New York Heart Association (NYHA) Class IV
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or corticosteroids)
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a pharmacologically pupil-dilated fundus examination performed by an ophthalmologist or another suitably qualified health care provider within the past 90 days prior to screening or in the period between screening and randomisation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (39):
- United States (12):
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Renton, Washington
- Canada (7):
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Concord, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Sarnia, Ontario
  - Novo Nordisk Investigational Site, Saint-Marc-des-Carrieres, Quebec
- Czechia (5):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Pardubice
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Rakovník
  - Novo Nordisk Investigational Site, Slaný
- Greece (2):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- Poland (6):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wierzchosławice
- Slovakia (5):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Moldava nad Bodvou
  - Novo Nordisk Investigational Site, Šahy
  - Novo Nordisk Investigational Site, Trenčín
- Slovenia (2):
  - Novo Nordisk Investigational Site, Koper
  - Novo Nordisk Investigational Site, Ljubljana

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Rosenstock J, Bajaj HS, Janež A, Silver R, Begtrup K, Hansen MV, Jia T, Goldenberg R. Once-Weekly Insulin for Type 2 Diabetes without Previous Insulin Treatment. PMID:32960514
- [Derived] Rosenstock J, Bajaj HS, Janez A, Silver R, Begtrup K, Hansen MV, Jia T, Goldenberg R; NN1436-4383 Investigators. Once-Weekly Insulin for Type 2 Diabetes without Previous Insulin Treatment. N Engl J Med. 2020 Nov 26;383(22):2107-2116. doi: 10.1056/NEJMoa2022474. Epub 2020 Sep 22. PMID 32960514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 49 sites in Canada (7), Czech Republic (9), Greece (5), Poland (6), Slovakia (6),Slovenia (2) and United States (14). One site in the United States screened, but didn't randomise any participant.
Pre-assignment Details: Insulin-naïve participants with Type 2 Diabetes (T2D) inadequately controlled on metformin with or without dipeptidyl peptidase 4 inhibitor (DPP4i) were randomized in a 1:1 manner to receive once weekly insulin 287 and once daily placebo or once weekly placebo and once daily insulin glargine subcutaneously (s.c).
Groups:
- Insulin 287: Participants were to receive once weekly s.c. injection of insulin 287 using PDS290 prefilled pen-injector at a starting dose of 70 units (U) and once daily placebo for 26 weeks. The insulin dose was then adjusted once weekly to reach the glycaemic target of 3.9-6.0 millimoles per liter (mmol/L) based on 3 pre-breakfast self-measured plasma glucose (SMPG) values measured on 2 previous days and on the day of the titration. If at least one pre-breakfast SMPG value was: < 3.0 mmol/L- dose reduced by 28 U, and 3.0-3.8- dose reduced by 14 U. Otherwise, the dose adjustment was based on the mean of SMPG values. If the mean was: 3.9-6.0 mmol/L- no adjustment; 6.1-7.0 mmol/L- dose increased by 14U, and >7.0 mmol/L- dose increased by 28U. All participants used metformin with or without DPP4i at the stable, pre-trial dose and at the same frequency unless due to safety concerns.
- Insulin Glargine: Participants were to receive once daily s.c injection of Insulin glargine using 10 ml vial and syringe at a starting dose of 10 U and once weekly placebo for 26 weeks. The insulin dose was then adjusted to reach the glycaemic target of 3.9-6.0 mmol/L based on 3 pre-breakfast SMPG values measured on 2 previous days and on the day of the titration. If at least one pre-breakfast SMPG value was: < 3.0 mmol/L- dose reduced by 4 U, and 3.0-3.8 dose reduced by 2 U. Otherwise, the dose adjustment was based on the mean of SMPG values. If the mean was: 3.9-6.0 mmol/L- no adjustment; 6.1-7.0 mmol/L- dose increased by 2 U, and >7.0 mmol/L- dose increased by 4 U. All participants used metformin with or without DPP4i at the stable, pre-trial dose and at the same frequency unless due to safety concerns.
Period: Overall Study
Arm/Group | Insulin 287 | Insulin Glargine
Started | 125 | 122
Completed | 122 | 119
Not Completed | 3 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin 287 | Insulin Glargine | Total
Number analyzed (Participants) | 125 | 122 | 247
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (8.2) | 59.4 (9.5) | 59.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 53 | 108
  Male | 70 | 69 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 115 | 116 | 231
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 5 | 12
  White | 109 | 113 | 222
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin (HbA1c) [Percentage Point (%-Point)]
Description: Change in HbA1c from baseline (week 0) to week 26 is presented. The endpoint was evaluated based on the data from on-treatment without ancillary treatment period, starting at the date of first dose of trial product until the follow-up visit, or the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin, or initiation of any diabetes treatment other than trial products and metformin +/- DPP4i, or increase of the dose of metformin or DPP4i.
Time Frame: From baseline (Visit 2) to week 26 (Visit 28)
Population: FAS included all randomised participants. "Number of Participants Analyzed" = Number of participants contributing to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage point of HbA1c
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 122 | 120
Percentage point of HbA1c | -1.33 (0.07) | -1.15 (0.07)
Statistical Analysis 1: Comparison: Insulin 287 vs Insulin Glargine; The response and change from baseline in response after 26 weeks are analysed using a linear mixed model for repeated measures (MMRM) with an unstructured covariance matrix and treatment, region, use of DPP-4 inhibitor and visit as fixed factors, and baseline response as covariate. Furthermore, the model includes the interaction between visit and all explanatory variables; Test type: Other; p = 0.0818, Mixed Models Analysis; Treatment difference = -0.18, 95% CI 2-sided [-0.38 to 0.02]

2. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose from baseline (week 0) to week 26 is presented. The endpoint was evaluated based on the data from on-treatment without ancillary treatment period, starting at the date of first dose of trial product until the follow-up visit, or the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin, or initiation of any diabetes treatment other than trial products and metformin +/- DPP4i, or increase of the dose of metformin or DPP4i.
Time Frame: From baseline (Visit 2) to week 26 (Visit 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/l
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 121 | 116
mmol/l | -3.20 (0.16) | -2.99 (0.16)

3. Secondary Outcome: 9-point Profile (Individual SMPG Values)
Description: Participants measured their plasma glucose (PG) levels using blood glucose meters (as plasma equivalent values of capillary whole blood glucose) at 9 time points (before breakfast, 90 minutes after the start of breakfast, before lunch, 90 minutes after the start of lunch, before dinner, 90 minutes after the start of dinner, at bedtime, at 4 am, before breakfast the following day). 9-point SMPG values after 26 weeks are presented. The endpoint was evaluated based on the data from on-treatment without ancillary treatment period, starting at the date of first dose of trial product until the follow-up visit, or the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin, or initiation of any diabetes treatment other than trial products and metformin +/- DPP4i, or increase of the dose of metformin or DPP4i.
Time Frame: Week 26 (Visit 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/l
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 125 | 122
mmol/l
  Before breakfast: number analyzed (Participants) | 109 | 108
  Before breakfast | 5.70 (0.19) | 6.19 (0.19)
  90 minutes after start of breakfast: number analyzed (Participants) | 103 | 107
  90 minutes after start of breakfast | 7.90 (0.19) | 8.51 (0.19)
  Before lunch: number analyzed (Participants) | 109 | 106
  Before lunch | 6.09 (0.19) | 6.19 (0.19)
  90 minutes after start of lunch: number analyzed (Participants) | 107 | 106
  90 minutes after start of lunch | 7.83 (0.19) | 8.50 (0.19)
  Before main evening meal: number analyzed (Participants) | 108 | 107
  Before main evening meal | 6.55 (0.19) | 6.96 (0.19)
  90 minutes after the start of main evening meal: number analyzed (Participants) | 106 | 104
  90 minutes after the start of main evening meal | 8.01 (0.19) | 8.47 (0.19)
  Before bedtime: number analyzed (Participants) | 104 | 105
  Before bedtime | 7.35 (0.19) | 7.87 (0.19)
  At 4:00 a.m.: number analyzed (Participants) | 101 | 102
  At 4:00 a.m. | 5.72 (0.19) | 5.98 (0.19)
  Before breakfast the following day: number analyzed (Participants) | 109 | 108
  Before breakfast the following day | 5.74 (0.19) | 6.05 (0.19)

4. Secondary Outcome: Change in Mean of the 9-point Profile, Defined as the Area Under the Profile Divided by Measurement Time
Description: Participants measured their PG levels using blood glucose meters at 9 time points (before breakfast, 90 minutes after the start of breakfast, before lunch, 90 minutes after the start of lunch, before dinner, 90 minutes after the start of dinner, at bedtime, at 4 am, before breakfast the following day). The endpoint was evaluated based on the data from on-treatment without ancillary treatment period, starting at the date of first dose of trial product until the follow-up visit, or the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin, or initiation of any diabetes treatment other than trial products and metformin +/- DPP4i, or increase of the dose of metformin or DPP4i.
Time Frame: From baseline (Visit 2) to week 26 (Visit 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/l
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 112 | 111
mmol/l | -2.70 (0.12) | -2.26 (0.12)

5. Secondary Outcome: Fluctuations of the 9-point Profile (Defined as the Integrated Absolute Distance From the Mean Profile Value Divided by Measurement Time).
Description: Participants measured their plasma glucose (PG) levels using blood glucose meters at 9 time points (before breakfast, 90 minutes after the start of breakfast, before lunch, 90 minutes after the start of lunch, before dinner, 90 minutes after the start of dinner, at bedtime, at 4 am, before breakfast the following day). Presented fluctuation in 9-point SMPG profile is the integrated absolute distance from the mean profile value divided by measurement time and is calculated using the trapezoidal method. The endpoint was evaluated based on the data from on-treatment without ancillary treatment period, starting at the date of first dose of trial product until the follow-up visit, or the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin, or initiation of any diabetes treatment other than trial products and metformin +/- DPP4i, or increase of the dose of metformin or DPP4i.
Time Frame: Week 26 (Visit 28)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/l
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 112 | 111
mmol/l | 0.92 [0.84 to 1.01] | 0.94 [0.86 to 1.03]

6. Secondary Outcome: Fasting C-peptide
Description: Fasting C-peptide at week 26 is presented. The endpoint was evaluated based on the data from on-treatment without ancillary treatment period, starting at the date of first dose of trial product until the follow-up visit, or the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin, or initiation of any diabetes treatment other than trial products and metformin +/- DPP4i, or increase of the dose of metformin or DPP4i.
Time Frame: At week 26 (Visit 28)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Nanomoles per liter (nmol/l)
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 115 | 112
Nanomoles per liter (nmol/l) | 0.44 [0.40 to 0.48] | 0.47 [0.43 to 0.51]

7. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to week 26 is presented. The endpoint was evaluated based on the data from on-treatment without ancillary treatment period, starting at the date of first dose of trial product until the follow-up visit, or the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin, or initiation of any diabetes treatment other than trial products and metformin +/- DPP4i, or increase of the dose of metformin or DPP4i.
Time Frame: From baseline (Visit 2) to week 26 (Visit 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilogram
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 122 | 119
Kilogram | 1.49 (0.36) | 1.56 (0.37)

8. Secondary Outcome: Weekly Dose of Insulin 287 and Weekly Dose of Insulin Glargine
Description: Weekly dose of insulin 287 and weekly dose of glargine at week 25 and week 26 are presented.The endpoint was evaluated based on the data from on-treatment without ancillary treatment period, starting at the date of first dose of trial product until the follow-up visit, or the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin, or initiation of any diabetes treatment other than trial products and metformin +/- DPP4i, or increase of the dose of metformin or DPP4i.
Time Frame: week 25 (Visit 27) and 26 (Visit 28)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units of Insulin
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 120 | 117
Units of Insulin | 229.06 [205.08 to 255.83] | 284.05 [253.97 to 317.71]

9. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial subject administered or using a medicinal product, whether or not considered related to the medicinal product or usage. A TEAE was defined as an event that had onset date (or increase in severity) during the on-treatment observation period. The endpoint was evaluated based on the data from on-treatment period, starting at the date of first dose of trial product, and ending at follow-up visit, or the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin.
Time Frame: From baseline (Visit 2) to week 31 (Visit 30)
Population: The safety analysis set (SAS) included all participants who received at least one dose of the investigational product or comparator.
Measure: Number; unit: Events
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 125 | 122
Events | 229 | 158

10. Secondary Outcome: Number of Hypoglycaemic Alert Episodes (Level 1) (≥3.0 and <3.9 mmol/L (≥54 and <70 mg/dL), Confirmed by BG Meter)
Description: Hypoglycaemia alert value (level 1) was defined as episodes that were sufficiently low for treatment with fast-acting carbohydrate and dose adjustment of glucose-lowering therapy with plasma glucose value of equal to or above (>=) 3.0 and less than (<) 3.9 mmol/L (>= 54 and < 70 mg/dL) confirmed by BG meter. Number of hypoglycaemic alert episodes (level 1) that occurred from week 0 to week 26 are presented.
Time Frame: From baseline (Visit 2) to week 26 (Visit 28)
Population: SAS included all participants who received at least one dose of the investigational product or comparator.
Measure: Number; unit: Episodes
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 125 | 122
Episodes | 358 | 145

11. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Clinically significant hypoglycaemic episodes (level 2) were defined as episodes that were sufficiently low to indicate serious, clinically important hypoglycaemia with plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL). Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. Number of clinically significant hypoglycaemic episodes (level 2), confirmed by blood glucose (BG) meter or severe hypoglycaemic episodes (level 3) that occurred from week 0 to week 26 are presented.
Time Frame: From baseline (Visit 2) to week 26 (Visit 28)
Population: SAS included all participants who received at least one dose of the investigational product or comparator.
Measure: Number; unit: Episodes
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 125 | 122
Episodes | 38 | 31

12. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3)
Description: Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. Number of severe hypoglycaemic episodes that occurred from week 0 to week 26 are presented.
Time Frame: From baseline (Visit 2) to week 26 (Visit 28)
Population: SAS included all participants who received at least one dose of the investigational product or comparator.
Measure: Number; unit: Episodes
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 125 | 122
Episodes | 1 | 0

13. Secondary Outcome: Change in Anti-insulin 287 Antibody Titres
Description: Samples from the insulin 287 arm of the study were analysed for anti-insulin 287 antibodies. Confirmed anti-insulin 287 antibody positive samples had an antibody titre value determined. The endpoint was evaluated based on the data from in-trial period, starting at randomisation, and ending at the last direct participant-site contact, or when participant withdrew their informed consent, or the last participant-investigator contact for participants lost to follow-up, or death.
Time Frame: From baseline (Visit 2) to week 31 (Visit 30)
Population: SAS included all participants who received at least one dose of the investigational product or comparator. Overall number of participants analysed = Number of participants contributing to the analysis.
Measure: Mean (Standard Deviation); unit: Antibody titers
Arm/Group | Insulin 287
Number analyzed (Participants) | 119
Antibody titers | 979.9 (3177.9)

14. Secondary Outcome: Change in Cross-reactive Anti-human Insulin Antibody Status (Positive/Negative)
Description: Anti-insulin 287 or glargine antibodies were classified as negative if % B/T was below a certain cut point. Samples positive for anti-insulin 287 or glargine antibodies were further tested for cross-reactivity to endogenous insulin. Samples not further tested are categorised as not applicable (NA). Unknown refers to samples with insufficient volume to perform analysis. The endpoint was evaluated based on the data from in-trial period, starting at randomisation, and ending at the last direct participant-site contact, or when participant withdrew their informed consent, or the last participant-investigator contact for participants lost to follow-up, or death.
Time Frame: From baseline (Visit 2) to week 31 (Visit 30)
Population: SAS included all participants who received at least one dose of the investigational product or comparator.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 125 | 122
Participants
  Week 0: Negative | 0 | 1
  Week 0: Positive | 0 | 0
  Week 0: Unknown | 1 | 9
  Week 0: Not Applicable | 124 | 112
  Week 31: number analyzed (Participants) | 120 | 115
  Week 31: Negative | 9 | 0
  Week 31: Positive | 86 | 26
  Week 31: Unknown | 0 | 0
  Week 31: Not Applicable | 25 | 89

15. Primary Outcome: Change in HbA1c [Millimoles/Mole (mmol/Mol)]
Description: as for outcome 1
Time Frame: From baseline (Visit 2) to week 26 (Visit 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/mol
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 122 | 120
mmol/mol | -14.51 (0.79) | -12.54 (0.80)
Statistical Analysis 1: Comparison: Insulin 287 vs Insulin Glargine; The response and change from baseline in response after 26 weeks are analysed using a linear MMRM with an unstructured covariance matrix and treatment, region, use of DPP-4 inhibitor and visit as fixed factors, and baseline response as covariate.Furthermore, the model includes the interaction between visit and all explanatory variables; Test type: Other; p = 0.0818, Mixed Models Analysis; Treatment difference = -1.97, 95% CI 2-sided [-4.19 to 0.25]

16. Secondary Outcome: Change in Anti-insulin 287 Antibody Level
Description: Change in anti-insulin 287 antibodies level is not assessed because change in anti-insulin 287 antibody titres is a more meaningful way of describing the change in antibody levels. The results for change in anti-insulin 287 antibody titres are reported as a separate endpoint.
Time Frame: From baseline (Visit 2) to week 31 (Visit 30)
Population: Change in anti-insulin 287 antibodies level is not assessed because change in anti-insulin 287 antibody titres is a more meaningful way of describing the change in antibody levels.
Arm/Group | Insulin 287 | Insulin Glargine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 0 to Week 31 Results are based on the SAS which included all participants who received at least one dose of Insulin 287 or Insulin glargine. The SAS included all participants who received at least one dose of the investigational product or comparator.
Description: A TEAE was defined as an event that had onset date (or increase in severity) during the on-treatment observation period. The endpoint was evaluated based on the data from on-treatment period, starting at the date of first dose of trial product, and ending at follow-up visit, or the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin.
Arm/Group | Insulin 287 | Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/122
Serious Adverse Events (participants affected / at risk) | 2/125 | 3/122
Other Adverse Events (participants affected / at risk) | 26/125 | 16/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin 287 (N=125) | Insulin Glargine (N=122)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Cerebral disorder (Nervous system disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Emphysematous pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin 287 (N=125) | Insulin Glargine (N=122)
Headache (Nervous system disorders) | 14 (31) | 3 (3)
Nasopharyngitis (Infections and infestations) | 10 (12) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT03751657/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT03751657/SAP_001.pdf